CLINICAL TRIAL: NCT01941472
Title: Transcutaneous pO2, Transcutaneous pCO2 and Central Venous SO2 Variations to Define Fluid Responsiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bin Du, Director of Medical ICU, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MICU2013-1
Record Dates: First submitted 2013-08-31; First posted 2013-09-13 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hypotension; Shock; Fluid Challenge; Fluid Responsiveness
MeSH Terms: conditions — Hypotension; Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Septic shock (Experimental): Adult patients (at least 18 years of age) with refractory hypotension secondary to sepsis who, at the discretion of treating physicians, required fluid challenge in the presence of invasive hemodynamic monitoring. Refractory hypotension was defined as need of vasopressors to maintain systolic blood pressure (SBP) no less than 90 mmHg despite adequate fluid resuscitation.
  Interventions: Other: fluid challenge

INTERVENTIONS:
Other: fluid challenge — A bag of 500ml of normal saline or 4% gelatin (Gelofusine, B. Braun Medical (Suzhou) Company Limited, Suzhou, China) is infused within 15 minutes using a bag pressurized to 300 mmHg. All other treatments, including maintenance fluids, dose of vasoactive agents and ventilator settings, remain unchanged during the study period.

SUMMARY:
Fluid challenge is often carried out in critical ill patients. Its responsiveness usually requires invasive monitoring. To use non-invasive methods is very tempting. Investigators hypothesize that transcutaneous pO2,transcutaneous pCO2 and Central Venous SO2 variations provide feasible estimation on fluid responsiveness in critical ill patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older ICU patients;
* Septic shock;
* Monitored with PICCO or Swan-Ganz catheter;
* The decision of fluid challenge made by the treating physician;

Exclusion Criteria:

* Evidence of fluid overload;
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MICU of Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu G, Huang H, Qin H, Du B. [Predictive value of central venous-to-arterial carbon dioxide partial pressure difference for fluid responsiveness in septic shock patients: a prospective clinical study]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2018 May;30(5):449-455. doi: 10.3760/cma.j.issn.2095-4352.2018.05.011. Chinese. PMID 29764550
- [Derived] Xu B, Yang X, Wang C, Jiang W, Weng L, Hu X, Peng J, Du B. Changes of central venous oxygen saturation define fluid responsiveness in patients with septic shock: A prospective observational study. J Crit Care. 2017 Apr;38:13-19. doi: 10.1016/j.jcrc.2016.09.030. Epub 2016 Oct 19. PMID 27829180

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Septic Shock
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Septic Shock
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 30
acute physiology and chronic health evaluation(APACHE) II score [Mean (Standard Deviation); unit: units on a scale] — acute physiology and chronic health evaluation(APACHE) II score can range from 0 to 71, with higher scores indicating more severe illness
  units on a scale | 27 (6)

OUTCOME MEASURES:

1. Primary Outcome: Fluid Responsiveness
Description: Increase in cardiac index ≥ 10% after fluid challenge
Time Frame: Immediately after fluid challenge, average 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Septic Shock
Number analyzed (Participants) | 40
Participants | 18

ADVERSE EVENTS:
Arm/Group | Septic Shock
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 40/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Septic Shock (N=40)
blood loss (Blood and lymphatic system disorders) | 40 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes